CLINICAL TRIAL: NCT01998971
Title: An Open-Label, Multicenter, Phase 1b Study of JNJ-54767414 (HuMax CD38) (Anti-CD38 Monoclonal Antibody) in Combination With Backbone Regimens for the Treatment of Subjects With Multiple Myeloma
Brief Title: A Study of JNJ-54767414 (HuMax CD38) (Anti-CD38 Monoclonal Antibody) in Combination With Backbone Treatments for the Treatment of Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR103015; 54767414MMY1001 (Other: Janssen Research & Development, LLC); 2013-003491-12 (EudraCT Number)
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Daratumumab; JNJ-54767414; Velcade-dexamethasone; Velcade-melphalan-prednisone; Velcade-thalidomide-dexamethasone; Pomalidomide-dexamethasone; Carfilzomib-dexamethasone; Carfilzomib-lenalidomide-dexamethasone; Anti-CD38 Monoclonal Antibody; Immunomodulatory drug; IMiD
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Bortezomib; pomalidomide; Dexamethasone; Melphalan; Prednisone; Thalidomide; Diphenhydramine; Acetaminophen; carfilzomib; Lenalidomide; montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (6):
- Daratumumab + VD (Experimental): Daratumumab will be administered with Velcade-dexamethasone (VD).
  Interventions: Drug: Daratumumab; Drug: Velcade; Drug: Dexamethasone; Drug: Diphenhydramine; Drug: Acetaminophen
- Daratumumab + VMP (Experimental): Daratumumab will be administered with Velcade-melphalan-prednisone (VMP).
  Interventions: Drug: Daratumumab; Drug: Velcade; Drug: Melphalan; Drug: Prednisone; Drug: Diphenhydramine; Drug: Acetaminophen
- Daratumumab + VTD (Experimental): Daratumumab will be administered with Velcade-thalidomide-dexamethasone (VTD).
  Interventions: Drug: Daratumumab; Drug: Velcade; Drug: Dexamethasone; Drug: Thalidomide; Drug: Diphenhydramine; Drug: Acetaminophen
- Daratumumab + Pom-dex (Experimental): Daratumumab will be administered with pomalidomide-dexamethasone (Pom-dex).
  Interventions: Drug: Daratumumab; Drug: Pomalidomide; Drug: Dexamethasone; Drug: Diphenhydramine; Drug: Acetaminophen
- Daratumumab + CFZ-dex (Experimental): Daratumumab will be administered with carfilzomib (CFZ)-dexamethasone (CFZ-dex) regimen.
  Interventions: Drug: Daratumumab; Drug: Dexamethasone; Drug: Diphenhydramine; Drug: Acetaminophen; Drug: Carfilzomib; Drug: Montelukast
- Daratumumab + KRd (Experimental): Daratumumab will be administered with carfilzomib- lenalidomide-dexamethasone (KRd) regimen.
  Interventions: Drug: Daratumumab; Drug: Dexamethasone; Drug: Diphenhydramine; Drug: Acetaminophen; Drug: Carfilzomib; Drug: Lenalidomide; Drug: Montelukast

INTERVENTIONS:
Drug: Daratumumab — Administered by either intravenous or subcutaneous infusions, in combination with the applicable backbone treatment.
Drug: Velcade — Administered subcutaneously in accordance with product labeling and local standards.
  Arms: Daratumumab + VD; Daratumumab + VMP; Daratumumab + VTD
Drug: Pomalidomide — Administered orally in accordance with product labeling and local standards.
  Arms: Daratumumab + Pom-dex
Drug: Dexamethasone — Administered intravenously or orally in accordance with product labeling and local standards.
  Arms: Daratumumab + CFZ-dex; Daratumumab + KRd; Daratumumab + Pom-dex; Daratumumab + VD; Daratumumab + VTD
Drug: Melphalan — Administered orally in accordance with product labeling and local standards.
  Arms: Daratumumab + VMP
Drug: Prednisone — Administered intravenously or orally in accordance with product labeling and local standards.
  Arms: Daratumumab + VMP
Drug: Thalidomide — Administered orally in accordance with product labeling and local standards.
  Arms: Daratumumab + VTD
Drug: Diphenhydramine — Administered in prophylactic doses intravenously (or equivalent) in accordance with product labeling and local standards.
Drug: Acetaminophen — Administered in prophylactic doses by mouth in accordance with product labeling and local standards.
Drug: Carfilzomib — Administered intravenously in accordance with product labeling and local standards.
  Arms: Daratumumab + CFZ-dex; Daratumumab + KRd
Drug: Lenalidomide — Administered orally in accordance with product labeling and local standards.
  Arms: Daratumumab + KRd
Drug: Montelukast — Administered intravenously or orally only with the first daratumumab dose in accordance with product labeling and local standards.
  Arms: Daratumumab + CFZ-dex; Daratumumab + KRd

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and dose regimen of daratumumab when administered in combination with various treatment regimens for the treatment of multiple myeloma.

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known) study to evaluate the safety, tolerability, and dose of daratumumab when administered in combination with various treatment regimens for different settings of multiple myeloma. The various treatment regimens to be combined with daratumumab in this study include Velcade-dexamethasone (VD), Velcade-melphalan-prednisone (VMP), Velcade-thalidomide-dexamethasone (VTD), pomalidomide-dexamethasone (Pom-dex), carfilzomib-dexamethasone (CFZ-dex) and carfilzomib-lenalidomide-dexamethasone (KRd). Approximately 250 patients (approximately 12 participants per VTD and VMP backbone treatment regimen, 6 for the VD regimen, up to 100 participants in the Pom-dex regimen, 80 for the CFZ-dex regimen [10 participants will receive a single-dose of daratumumab and the remaining participants will receive a split-dose of daratumumab], and up to 40 for the KRd regimen) will be enrolled in this study. The study will consist of screening, treatment, and follow-up phases. Treatment will extend to either the planned treatment duration for a maximum of 1 year (in Velcade-dexamethasone, Velcade-melphalan-prednisone, Velcade-thalidomide-dexamethasone regimens and KRd regimens), or in the Pom-dex and CFZ-dex regimens, until disease progression, unacceptable toxicity, or until the end of study. Follow-up will continue until the study ends (approximately 25 months after the last patient receives the first dose of daratumumab). Serial pharmacokinetic (study of what a drug does to the body) blood samples will be collected. Clinical efficacy outcomes and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of symptomatic multiple myeloma and measurable secretory disease
* For carfilzomib-lenalidomide-dexamethasone (KRd) regimen: newly diagnosed myeloma. For carfilzomib-dexamethasone (CFZ-dex) regimen: relapsed or refractory disease
* Eastern Cooperative Oncology Group performance status score of 0, 1, or 2
* Pretreatment clinical laboratory values must meet protocol-defined parameters during the screening phase

Exclusion Criteria:

* Previously received daratumumab or other anti-CD38 therapies
* Diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance, smoldering multiple myeloma, Waldenström's disease, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions
* Peripheral neuropathy or neuropathic pain Grade 2 or higher
* Prior or concurrent invasive malignancy (other than multiple myeloma) within 5 years of study start
* Exhibiting clinical signs of meningeal involvement of multiple myeloma
* Known chronic obstructive pulmonary disease, persistent asthma, or a history of asthma within 2 years
* Seropositive for human immunodeficiency virus, hepatitis B, or hepatitis C
* Any concurrent medical or psychiatric condition or disease that is likely to interfere with the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in this study
* Clinically significant cardiac disease
* Plasma cell leukemia or POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-02-18 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Number of participants affected by adverse events by MedDRA system organ class (SOC) and Preferred term (PT) | Up to 30 days after the last dose of study medication
Number of participants affected by dose-limiting toxicities | Up to 30 days after the last dose of study medication

SECONDARY OUTCOMES:
Maximum observed concentration of daratumumab | Up to post-treatment visit Week 9
Number of participants with generation of antibodies to daratumumab | Up to post-treatment visit Week 9
Complete response rate | Up to 25 months after last patient receives first dose of study drug
Overall response rate | Up to 25 months after last patient receives first dose of study drug
Duration of response | Up to 25 months after last patient receives first dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (22):
- United States (10):
  - Duarte, California
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - New York, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Philadelphia, Pennsylvania
  - Dallas, Texas
- France (6):
  - Lille
  - Nantes
  - Paris
  - Pessac
  - Toulouse
  - Tours
- Spain (6):
  - Badalona
  - Barcelona
  - Madrid
  - Pamplona
  - Salamanca
  - Valencia

REFERENCES:
- [Derived] Moreau P, Chari A, Oriol A, Martinez-Lopez J, Haenel M, Touzeau C, Ailawadhi S, Besemer B, de la Rubia Comos J, Encinas C, Mateos MV, Salwender H, Rodriguez-Otero P, Hulin C, Karlin L, Sureda Balari A, Bargay J, Benboubker L, Rosinol L, Tarantolo S, Terebelo H, Yang S, Wang J, Nnane I, Qi M, Kosh M, Delioukina M, Goldschmidt H. Daratumumab, carfilzomib, and dexamethasone in relapsed or refractory myeloma: final analysis of PLEIADES and EQUULEUS. Blood Cancer J. 2023 Mar 7;13(1):33. doi: 10.1038/s41408-023-00805-x. No abstract available. PMID 36882409
- [Derived] He J, Berringer H, Heeg B, Ruan H, Kampfenkel T, Dwarakanathan HR, Johnston S, Mendes J, Lam A, Bathija S, Mackay EK. Indirect Treatment Comparison of Daratumumab, Pomalidomide, and Dexamethasone Versus Standard of Care in Patients with Difficult-to-Treat Relapsed/Refractory Multiple Myeloma. Adv Ther. 2022 Sep;39(9):4230-4249. doi: 10.1007/s12325-022-02226-x. Epub 2022 Jul 22. PMID 35876974
- [Derived] Leleu X, Beksac M, Chou T, Dimopoulos M, Yoon SS, Prince HM, Pour L, Shelekhova T, Chari A, Khurana M, Zhang J, Obreja M, Qi M, Oriol A, Siegel D. Efficacy and safety of weekly carfilzomib (70 mg/m2), dexamethasone, and daratumumab (KdD70) is comparable to twice-weekly KdD56 while being a more convenient dosing option: a cross-study comparison of the CANDOR and EQUULEUS studies. Leuk Lymphoma. 2021 Feb;62(2):358-367. doi: 10.1080/10428194.2020.1832672. Epub 2020 Oct 28. PMID 33112184
- [Derived] Xu XS, Moreau P, Usmani SZ, Lonial S, Jakubowiak A, Oriol A, Krishnan A, Blade J, Luo M, Sun YN, Zhou H, Nnane I, Deraedt W, Qi M, Ukropec J, Clemens PL. Split First Dose Administration of Intravenous Daratumumab for the Treatment of Multiple Myeloma (MM): Clinical and Population Pharmacokinetic Analyses. Adv Ther. 2020 Apr;37(4):1464-1478. doi: 10.1007/s12325-020-01247-8. Epub 2020 Feb 20. PMID 32078124
- [Derived] Chari A, Martinez-Lopez J, Mateos MV, Blade J, Benboubker L, Oriol A, Arnulf B, Rodriguez-Otero P, Pineiro L, Jakubowiak A, de Boer C, Wang J, Clemens PL, Ukropec J, Schecter J, Lonial S, Moreau P. Daratumumab plus carfilzomib and dexamethasone in patients with relapsed or refractory multiple myeloma. Blood. 2019 Aug 1;134(5):421-431. doi: 10.1182/blood.2019000722. Epub 2019 May 21. PMID 31113777
- [Derived] Chari A, Suvannasankha A, Fay JW, Arnulf B, Kaufman JL, Ifthikharuddin JJ, Weiss BM, Krishnan A, Lentzsch S, Comenzo R, Wang J, Nottage K, Chiu C, Khokhar NZ, Ahmadi T, Lonial S. Daratumumab plus pomalidomide and dexamethasone in relapsed and/or refractory multiple myeloma. Blood. 2017 Aug 24;130(8):974-981. doi: 10.1182/blood-2017-05-785246. Epub 2017 Jun 21. PMID 28637662